CLINICAL TRIAL: NCT02651168
Title: Predictors of Treatment Response to Aflibercept and Aqueous Cytokine Levels in Patients With Persistent Diabetic Macular Edema Following Treatment With Ranibizumab: An Interventional Prospective Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol B SMH Aflibercept
Record Dates: First submitted 2016-01-07; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; Ocular Cytokines; aflibercept; ranibizumab
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- aflibercept (Other): aflibercept treatment aflibercept, 40 mg/mL Solution for Intravitreal Injection
  Interventions: Biological: aflibercept

INTERVENTIONS:
Biological: aflibercept — EYLEA (aflibercept, solution for intravitreal injection) is a recombinant fusion protein consisting of portions of human Vascular Endothelial Growth Factor (VEGF) receptor 1 and 2 extracellular domains fused to the Fc portion of human IgG1 and formulated as an iso-osmotic solution for intravitreal administration. Aflibercept is produced in Chinese hamster ovary (CHO) K1 cells by recombinant DNA technology.
  Other Names: Eylea

SUMMARY:
Diabetic macular edema refers to swelling (fluid accumulation) in the center of the retina. The retina is like the film of a camera and is located in the back of the eye. This condition can develop in diabetics where swelling results from leaking of fluid from the blood vessels of the eye, into the center of the retina, the macula. If left untreated, this can affect central.

The current standard treatment for diabetic macular edema includes medications injected directly into the eye (intravitreal injections) and laser eye treatment. The drugs that are injected directly into the eye are known as anti-VEGF agents which help to reduce the leaking. This includes bevacizumab (Avastin®) and ranibizumab (Lucentis®).

However, some patients do not respond well to these anti-VEGF treatments and will be given the option of switching to an another newer anti-VEGF medication, called aflibercept (Eylea®) that is approved to treat DME. A recent large study has demonstrated that aflibercept was as efficacious as other anti-VEGF therapies listed above and was even superior in patients with worse vision (Diabetic Retinopathy Clinical Research Network, Wells JA, Glassman AR, et al. Aflibercept, Bevacizumab, or Ranibizumab for Diabetic Macular Edema. N Engl J Med. 2015:150218140025008-150218140025008).

The purpose of this study is to determine what factors affect the treatment response to aflibercept (amount of swelling reduction) for patients with diabetic macular edema, who were previously unresponsive to ranibizumab injections.

ELIGIBILITY:
Inclusion Criteria

* Male or female aged 18 years or above
* Presence of Non Proliferative Diabetic Retinopathy (NPDR)
* Prior treatment with ≥ 6 intravitreal ranibizumab injections but no treatment in the last 4 weeks and less than 10% improvement in Central Macular Thickness on OCT scan and less than 1 line improvement in vision from baseline and less than 10% reduction in macular volume with Snellan Acuity 20/40 to 20/400
* Patients with DME with central macular thickness of 310μm or more on SD-OCT (cirrus)
* Subjects with Type I or II diabetes mellitis
* Willing and able to provide informed consent for participation in the study

Exclusion Criteria

* Proliferative diabetic retinopathy in the study eye or PRP within the last 12 months or anticipated PRP in the next 6 months
* Uncontrolled glaucoma
* History of intraocular surgery within 3 months in the study eye
* History of vitrectomy surgery
* Laser treatment within 3 months of study eye
* Vitreomacular traction, epiretinal membrane or any other maculopathy in the study eye
* Prior intravitreal injection within the past 6 months
* Known allergy to the study drug or fluorescein
* History of stroke or AMI within 6 months of enrolment
* Patients receiving dialysis for renal failure
* Patients currently on systemic immunosuppression
* Patients on two or more class of medication for glaucoma in study eye
* Patients with tuberculosis
* Patients who are pregnant.
* Unwilling or unable to follow or comply with all study related procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change in cytokine levels (picograms per mL) in patients with DME who were previously non-responders to ranibizumab (non-responders) between baseline aflibercept injection. | 1month, 2 months, 3 months

SECONDARY OUTCOMES:
Relation of baseline aqueous cytokine levels in patients with DME who were previously non-responders to ranibizumab (non-responders) to baseline Snellen BCVA in response to aflibercept | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev Muni, MD, Principal Investigator — St. Michael's Hospital Eye Clinic, Toronto, Ontario, Canada, M5C2T2